CLINICAL TRIAL: NCT03394274
Title: Restrictive Versus Liberal Transfusion for Elective Major Surgery and Perioperative Outcomes: Mortality, Morbidity and Requirement of Postoperative Blood Transfusion
Brief Title: Restrictive Versus Liberal Transfusion, Major Surgeries
Acronym: transfusion
Status: Completed | Type: Observational
Sponsor: Leyla Kılınc (Other)
Responsible Party: Sponsor-Investigator, Leyla Kılınc, medical doctor, anesthesiology specialist, Sisli Hamidiye Etfal Training and Research Hospital
Organization: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Other Study IDs: 814
Record Dates: First submitted 2017-11-27; First posted 2018-01-09 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Transfusion Related Complication
Keywords: transfusion; liberal; restrictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transfusion: Patients (n:892) were enrolled who underwent elective major surgery between the 01/01/2016-31/12/2016, and over the age of 18 years. They separated subgroups as restrictive and liberal blood transfusion groups
  Interventions: Other: restrictive and liberal transfusion

INTERVENTIONS:
Other: restrictive and liberal transfusion — hemoglobin threshold value was accepted 8g/dl. restrictive blood transfusion group was defined that if perioperative transfusion was started equal or under hemoglobin level 8 g / dL. Liberal blood transfusion group was defined as perioperative transfusion was started over hemoglobin level 8 g / dL .

SUMMARY:
Investigators aimed to compare the restrictive and liberal blood transfusion methods applied in major surgical operations performed in Anesthesiology and Reanimation Clinic and investigate their effects on postoperative transfusion needs, morbidity and mortality.

DETAILED DESCRIPTION:
The test subjects consisted of 892 patients, who belong to ASA (American society of Anesthesiology) I -IV groups, underwent elective major surgery between the 01/01/2016-31/12/2016, and are over the age of 18 years. The demographic data (Age, sex, ASA (American society of Anesthesiology) scors, surgery type) were also recorded. we evaluated the value of Hemoglobin, platelet, APTT (activated partial thromboplastin time), INR (international normalized ratio) preoperatively and postoperatively. In this study, restrictive and liberal blood transfusion groups were investigated.restrictive and liberal transfusion hemoglobin threshold value respectively before perioperative transfusion was 8 g / dL. were defined as restrictive blood transfusion group and perioperative transfusion was over 8 g / dL were defined as liberal blood transfusion group. Adverse events (tachycardia, hypotension, the value of lactate and metabolic acidosis). Postoperatively, the amount of postoperative transfusion unit, duration of hospital stay, requirement of intensive care unit and mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old patients,
* ASA I-II-III-IV,
* Major surgeries ( Intra-abdominal, intracranial, head and neck malignancy surgery, femur and vertebra surgery)

Exclusion Criteria:

* Emergency operation,
* Cardiovascular surgery,
* ASA V-VI
* Under 18 years old patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 years old patients, ASA I-II-III-IV, major surgeries ( Intraabdominal, intracranial, head and neck malignanacy surgery, femur and vertebra surgery) were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 892 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Restrictive or Liberal transfusion | 52 weeks
  It is determined how many units of RBC (red blood cell ) used during major operations at the hospital in liberal transfusion group or restrictive transfusion group.

SECONDARY OUTCOMES:
Mortality | 52 weeks
  Survival ratios between the restrictive transfusion group and the liberal transfusion group are compared.
Postoperative transfusion requirement | 52 Weeks
  The requirement of postoperative blood transfusion between the restrictive transfusion group and the liberal transfusion group is determined.
The Need of ICU | 52 Weeks
  The need of ICU between the restrictive transfusion group and the liberal transfusion group of patients is determined.
Postoperative Duration of Stay in Hospital of patients | 52 Weeks
  The postoperative duration of stay in hospital of patients between the restrictive transfusion group and the liberal transfusion group are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health sciences,sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Meier J, Filipescu D, Kozek-Langenecker S, Llau Pitarch J, Mallett S, Martus P, Matot I; ETPOS collaborators. Intraoperative transfusion practices in Europe. Br J Anaesth. 2016 Feb;116(2):255-61. doi: 10.1093/bja/aev456. PMID 26787795